CLINICAL TRIAL: NCT02609152
Title: Effect of a Continuous Infusion of Esmolol on Stroke Volume in Patients With Hyperdynamic Vasoplegic Septic Shock: a Multicentre, Randomized, Double-blind Trial
Brief Title: Effect of a Continuous Infusion of Esmolol on Stroke Volume in Patients With Hyperdynamic Vasoplegic Septic Shock
Acronym: BétaSep
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: logistical difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOCAL/2014/ML-01; 2015-000895-90 (EudraCT Number)
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Shock, Septic
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous perfusion of esmolol (Experimental): Intervention: Drug: Continuous perfusion of esmolol
  Interventions: Drug: Continuous perfusion of esmolol
- Continuous perfusion of saline (Placebo Comparator): Intervention: Continuous perfusion of saline
  Interventions: Drug: Continuous perfusion of saline

INTERVENTIONS:
Drug: Continuous perfusion of esmolol — In the experimental arm of the study, a continuous perfusion of esmolol will be performed. This infusion starts at 5 ml / h with an increase of 5 ml / hr every 10 minutes to obtain a 15% decrease in heart rate. The infusion will be reduced by 5 ml / h every 5 minutes if the cardiac rate is less than 90 beats per minute and stopped if it is less than 70 beats per minute. At H4, the doctor in charge is free to gradually continue or stop the infusion.
  Arms: Continuous perfusion of esmolol
Drug: Continuous perfusion of saline — In the control arm of the study, a continuous infusion of normal saline will be performed. This infusion starts at 5 ml / h with an increase of 5 ml / hr every 10 minutes to obtain a 15% decrease in heart rate. The infusion will be reduced by 5 ml / h every 5 minutes if the cardiac rate is less than 90 beats per minute and stopped if it is less than 70 beats per minute. A H4, the doctor in charge is free to gradually continue or stop the infusion.
  Arms: Continuous perfusion of saline

SUMMARY:
The main objective of this study is to evaluate the effectiveness of the administration of a short acting beta-blocker in terms of effective increase in stroke volume (at least 15%) after 4 hours initiation of therapy in septic shock in patients with a hyperkinetic profile after 12-24 hours of care.

This research seeks to demonstrate that the proportion of patients with an increase in the systolic ejection superior or equal to 15% (relative to baseline) at four hours is different between the two arms of the study: (1) an experimental arm where patients receive an esmolol infusion according to a predetermined procedure and (2) a control arm where patients receive a saline infusion according to a predetermined procedure.

DETAILED DESCRIPTION:
The secondary objectives are to compare the following items between the two arms of the study:

A. Central venous oxygen saturation at 4 hours (H4)

B. Changes in plasma concentration of lactates between H0 and H4

C. Changes in the tissue oxygen saturation between H0 and H4

D. Changes in echocardiographic parameters of systolic function of the left ventricle (LV) and right ventricle (RV), as well as diastolic LV function between H0 and H4

E. Vascular Filling volume during the study period

F. Kidney function: urine output and creatinine changes between H0 and H4

G. The required vasopressor time between H0 and H4

H. Use of positive inotropic agents

I. The inflammatory response via the analysis of HLA-DR between H0 and H4 and M1 / M2 responses at H4

J. The duration of ICU stay, mortality, morbidity in terms of organ failures

ELIGIBILITY:
Inclusion Criteria:

* The patient or his/her representative was informed about the implementation of the study, its objectives, constraints and patient rights or emergency consent
* The patient or his/her representative must haven given free and informed consent and signed the consent or emergency consent
* The patient must be affiliated with or the recipient of a health insurance plan
* Septic shock criteria: shock for which the suspected or proven starting point is an infection requiring vasopressors after adequate fluid resuscitation that started within the past 24 to 72 hours
* Precharge independence criteria obtained: i.e. pulsed pressure variation <13% or variation in ejection volume <10% or variation in the cardiac index after passive lift leg <10% or central venous pressure between 8 and 12 mmHg.
* Antibiotic treatment in progress
* Prescription ongoing vasopressor for 24 to 72 hours.
* Sinus rhythm
* Heart rate > 100 beats per minute
* Cardiac Index measured by thermodilution greater than 4.0 l / min / m^2
* Central venous oxygen saturation > 80% without positive inotropics such as dobutamine or isoproterenol (continuously taken or measured via central venous line in superior vena cava territory) on two successive samples in 12 hours
* Monitoring of stroke volume (invasive, semi-invasive or ultrasound)

Exclusion Criteria:

* The patient is participating in another study
* The patient has participated in another study in the last 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under any kind of guardianship
* The patient is under judicial protection
* The patient or his/her representative refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for a treatment used in this study
* Cardiac index < 4.0 l / min / m^2
* Need to introduce a positive inotropic agent (as determined by the physician in charge of the patient)
* Contraindications to the use of esmolol: Severe sinus bradycardia (less than 50 beats per minute); Sinus pathologies, severe disorders of atrioventricular conduction (without pacemaker), atrioventricular blocks of second and third degree; Cardiogenic shock; Severe hypotension; Decompensated heart failure; Untreated pheochromocytoma; Pulmonary hypertension; Acute asthma attack; chronic obstructive pulmonary disease; peripheral arterial disease; Metabolic acidosis; Known hypersensitivity to esmolol.
* Patient with kidney failure (RIFLE Stage L)
* Chronic treatment with beta blocker
* Patient with ultrasound assessment of left ventricular ejection fraction < 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Is stroke volume increased ≥ 15% as compared to baseline? | 4 hours

SECONDARY OUTCOMES:
The time spent with a central venous oxygen saturation between 70% and 80% (minutes) | 4 hours
Evolution of blood lactate between H0 and H4 | 4 hours
Changes in tissue oxygen saturation compared to baseline | 4 hours
Ejection fraction of the left ventricle drops below 40% between H0 and H4? yes/no | 4 hours
the change (in %) of the systolic S wave on the tissue doppler at the mitral annulus relative to baseline | 4 hours
Change (%) in the sub aortic time-speed integral relative to baseline | 4 hours
Absolute values of the E wave | baseline (hour 0)
Absolute values of the E wave | 4 hours
Absolute values of the E' wave | baseline (hour 0)
Absolute values of the E' wave | 4 hours
Absolute value of the ratio E/A on pulsed Doppler at the mitral annulus | baseline (hour 0)
Absolute value of the ratio E/A on pulsed Doppler at the mitral annulus | 4 hours
Absolute Value of the ratio E/E ' one tissue Doppler at the mitral annulus | baseline (hour 0)
Absolute Value of the ratio E/E ' one tissue Doppler at the mitral annulus | 4 hours
Right ventricular systolic function | baseline (hour 0)
Right ventricular systolic function | 4 hours
right ventricle / left ventricle diameter ratio | baseline (hour 0)
right ventricle / left ventricle diameter ratio | 4 hours
Vascular filling volume (ml) | 4 hours
Diuresis (ml/kg/h) | collected between hours 0 and 4
Change in creatinine relative to baseline (µmol/L) | 4 hours
Required duration of vasopressors (min) | 4 hours
Use of positive ionotropic agents? yes/no | 4 hours
Percentage variation o, inflammatory cytokines (tissue necrosis factor) with respect to baseline values | 4 hours
Percentage variation o, inflammatory cytokines (interleukin 1) with respect to baseline values | 4 hours
Percentage variation o, inflammatory cytokines (interleukin 10) with respect to baseline values | 4 hours
Percentage change in the expression of the human leukocyte antigen-DR gene with respect to baseline | 4 hours
Length of stay in the intensive care unit (days) | Expected maximum of 28 days
  The maximum observed length of stay in the intensive care unit (days) = Dmax
Number of days free of organ failure | Dmax +1 (Dmax has an expected maximum of 28 days)
Mortality | Dmax +1 (Dmax has an expected maximum of 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Leone, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - APHM - Hôpital Nord, Marseille
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes